CLINICAL TRIAL: NCT03470610
Title: Administration of Vaginal and Rectal Progesterone During Frozen Embryo Transfer Cycles
Brief Title: Administration of Vaginal and Rectal Progesterone During FET Cycles
Status: Completed | Type: Observational
Sponsor: Thor Haahr (Other)
Responsible Party: Sponsor-Investigator, Thor Haahr, Professor, Regionshospitalet Viborg, Skive
Organization: Regionshospitalet Viborg, Skive (Other)
Other Study IDs: Progesterone03
Record Dates: First submitted 2018-03-12; First posted 2018-03-20 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Infertility
Keywords: Progesterone; HRT; frozen embryo transfer
MeSH Terms: conditions — Infertility | interventions — Progesterone; Estradiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Progesterone — 6 mg estradiol and vaginal and rectal progesterone
  Other Names: estradiol

SUMMARY:
Observational study of reproductive outcome after frozen embryo transfer in HRT with vaginal and rectal progesterone.

DETAILED DESCRIPTION:
Cohort of patients treated with autologous blastocyst at the Fertility clinic Skive Regional Hospital in HRT cycle. Estradiol stimulation started on second cycle day and on day 12 - 20 vaginal and rectal progesterone is added. Blastocyst transfer on 6th progesterone treatment day. Serum progesterone and hCG measurement 9 or 11 days after embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Frozen embryo transfer cycles in HRT cycles

Exclusion Criteria:

* Donor frozen embryo transfer

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Autologuos spare embryos from previous IVF/ICSI cycles.
Sampling Method: Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy | 4 month
  gestational week 12

SECONDARY OUTCOMES:
pregnancy rate | 4 month
  positive hCG
Pregnancy loss | 4 month
  pregnancy loss before week 7

CONTACTS AND LOCATIONS:
Overall Officials: Peter Humaidan, DMsc, Study Chair — Fertility Clinic Skive
Locations (1):
- Fertility Clinic Regional Hospital Skive, Skive, Denmark

IPD SHARING:
Plan to Share IPD: No